CLINICAL TRIAL: NCT04868344
Title: An Open-Label, Dose-Finding, Phase I Study in Solid Tumors.
Brief Title: A Study of MRG003 in Patients With Advanced Solid Tumors
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Shanghai Miracogen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: MRG003-001
Record Dates: First submitted 2021-04-29; First posted 2021-04-30 (Actual); Last update posted 2021-04-30 (Actual); Status verified 2021-04

CONDITIONS: Advanced Solid Tumors
Keywords: MRG003; Antibody Drug Conjugate (ADC); Solid tumors

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MRG003 (Experimental): Phase Ia: MRG003 will be administrated by an IV infusion of escalating doses (0.1, 0.3, 0.6, 1.0, 2.0, 2.5, 3.0 mg/kg) on Day 1 of every 3 weeks (Q3W); Phase Ib: MRG003 will be administrated by an IV infusion of MTD/RP2D.
  Interventions: Drug: MRG003

INTERVENTIONS:
Drug: MRG003 — Administered intravenously

SUMMARY:
The objective of this study is to assess the safety, efficacy, and pharmacokinetics of MRG003, as well as immunogenicity as defined by the incidence of anti-drug antibody (ADA) of MRG003 in patients with advanced solid tumors, including colorectal cancer, squamous cell carcinoma of head and neck, and nasopharyngeal carcinoma.

DETAILED DESCRIPTION:
This study consists of two parts: Phase Ia dose escalation and Phase Ib dose expansion. The objective of Phase Ia is to determine MTD or RP2D, and Phase Ib is conducted to evaluate efficacy of MRG003 in patients with advanced colorectal cancer, squamous cell carcinoma of head and neck (SCCHN), and nasopharyngeal carcinoma.

ELIGIBILITY:
Inclusion Criteria:

* Willing to sign the ICF and follow the requirements specified in the protocol.
* Age: ≥18 years and ≤75 years, both genders
* Expected survival time≥12 weeks
* Phase Ia: Patients with histologically and cytologically confirmed advanced or metastatic solid tumor
* Phase Ib: Patients with histologically and cytologically confirmed EGFR-positive advanced or metastatic colorectal cancer, squamous cell carcinoma of head and neck, and nasopharyngeal carcinoma
* Subjects must have measurable lesions according to the response Evaluation Criteria In Solid Tumors（RECIST v1.1）
* ECOG performance score 0 or 1
* Acceptable liver, renal, and hematologic function
* Patients with childbearing potential must use effective contraception during the treatment and for 6 months after the last dose of treatment

Exclusion Criteria:

* History of hypersensitivity to any component of the investigational product
* Presence of central nervous system metastasis
* Prior history of other primary malignancies
* Known history of clinically significant hepatic diseases
* Evidence of active infection of human immunodeficiency virus (HIV)
* History of ophthalmic abnormalities
* Any severe or uncontrolled systemic disease judged by the investigator
* Patients with poorly controlled heart diseases
* Received radiotherapy, chemotherapy, biotherapy, immunotherapy or other anti-tumor drugs within 4 weeks prior to the first dose of study treatment
* Major surgery or surgical therapy for any cause within 4 weeks prior to the first dose of investigational drug
* Planned surgery or surgery is the best interest of patients as determined by investigator
* History of severe skin disease requiring interruption of previous EGFR targeted therapy; or chronic skin disease requiring oral or intravenous therapy
* Active concomitant diseases that might increase risks of toxicity
* Pregnancy, or breast feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 61 (Actual)
Dates: Start 2018-05-09 (Actual); Primary Completion 2021-03-29 (Actual); Study Completion 2021-03-29 (Actual)

PRIMARY OUTCOMES:
Dose Limiting Toxicity (DLT) - Phase Ia | First cycle (21 days)
  DLT is assessed on Day 21 (Day 1 to 21) of the first dose administration.
Objective Response Rate (ORR) - Phase Ib | Baseline to study completion (up to 24 weeks)
  ORR was defined as the proportions of subjects with a complete response (CR) and partial response (PR). ORR will be assessed by investigator according to RECIST v1.1.

SECONDARY OUTCOMES:
PK parameter for MRG003: Maximum Drug Concentration (Cmax) | Baseline to study completion (up to 24 weeks)
  Cmax will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for MRG003: Area Under the Curve Up to the Last Validated Measurable Plasma Concentration (AUClast) | Baseline to study completion (up to 24 weeks)
  AUClast will be derived from the PK blood samples collected and will be summarized with descriptive statics.
PK parameter for total antibody (TAb): Cmax | Baseline to study completion (up to 24 weeks)
  Cmax will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for TAb: AUClast | Baseline to study completion (up to 24 weeks)
  AUClast will be derived from the PK blood samples collected and will be summarized with descriptive statics.
PK parameter for Monomethyl Auristatin E (MMAE): Cmax | Baseline to study completion (up to 24 weeks)
  Cmax will be derived from the PK blood samples collected and will be summarized with descriptive statistics.
PK parameter for MMAE: AUClast | Baseline to study completion (up to 24 weeks)
  AUClast will be derived from the PK blood samples collected and will be summarized with descriptive statics.
Immunogenicity | Baseline to study completion (up to 24 weeks)
  Blood samples for anti-drug antibody (ADA) analysis will be collected each time according to the pre-defined timepoints.
Progression Free Survival (PFS) - Phase Ib only | Baseline to study completion (up to 24 weeks)
  PFS was defined as the duration from the start of treatment to the onset of tumor progression or death of any cause.
Duration of Response (DoR) - Phase Ib only | Baseline to study completion (up to 24 weeks)
  DOR was defined as the duration from the initial recording of objective disease response to the first onset of tumor progression, or death of any cause.
Overall Survival (OS) - Phase Ib only | Baseline to study completion (up to 24 weeks)
  OS was defined as the duration from the start of treatment to death of any cause.
Incidence of Adverse Events (AEs) | Baseline to 30 days after the last dose of study treatment
  Incidence of AEs and serious adverse events (SAEs) will be assessed based on NCI-CTCAE v5.0

CONTACTS AND LOCATIONS:
Overall Officials: Ruihua Xu, M.D., Principal Investigator — Sun Yat-sen University
Locations (1):
- Sun Yat-sen University Cancer Center, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qiu MZ, Zhang Y, Guo Y, Guo W, Nian W, Liao W, Xu Z, Zhang W, Zhao HY, Wei X, Xue L, Tang W, Wu Y, Ren G, Wang L, Xi J, Jin Y, Li H, Hu C, Xu RH. Evaluation of Safety of Treatment With Anti-Epidermal Growth Factor Receptor Antibody Drug Conjugate MRG003 in Patients With Advanced Solid Tumors: A Phase 1 Nonrandomized Clinical Trial. JAMA Oncol. 2022 Jul 1;8(7):1042-1046. doi: 10.1001/jamaoncol.2022.0503. PMID 35511148